CLINICAL TRIAL: NCT05062226
Title: Evaluating the Tolerance, Safety and Acceptability of GMP-based Protein Substitutes for the Dietary Management of Phenylketonuria and Tyrosinaemia in Children and Adults: a Case Study Series
Brief Title: GMP Case Studies of Tolerance, Safety and Acceptability in PKU and TYR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nutricia UK Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: GMP2020
Record Dates: First submitted 2021-09-06; First posted 2021-09-30 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: PKU; Tyrosinemias
Keywords: PKU; TYR
MeSH Terms: conditions — Tyrosinemias

STUDY DESIGN:
Intervention Model Description: 15 patients per product will be included in the case studies for a total of 45 patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GMP-based products (Experimental): GMP-based nutritional protein substitutes for the dietary management of PKU and TYR
  Interventions: Dietary Supplement: PKU/TYR GMP Protein Substitute

INTERVENTIONS:
Dietary Supplement: PKU/TYR GMP Protein Substitute — After a 1-day baseline period during which patients will consume their usual protein substitute, each patient will receive one the case study product for 4 weeks (28 days).

SUMMARY:
Three new protein substitutes have been developed to help with compliance in PKU and TYR patients, which are powdered protein substitutes, low in Phe and, low in Phe and Tyr respectively, with a mixed balance of glycomacropeptide (GMP), essential and non-essential amino acids, carbohydrates, fats and micronutrients for the dietary management of PKU and TYR.

This series of case-studies will evaluate the acceptability, compliance, gastrointestinal tolerance and safety of the three GMP-based products for PKU and TYR in 45 patients with PKU and TYR, in both adults and children over 3 years (15 patients per product). The case study will last 29 days in total, including a 1-day baseline period followed by a 28-day intervention period. The case studies will be conducted across multiple specialist metabolic centres in the UK, to meet the UK ACBS and GMS requirements for acceptability studies. A series of case studies is undertaken due to the rarity of these conditions and the difficulty in recruiting these patients to trials.

DETAILED DESCRIPTION:
Phenylketonuria (PKU) and Tyrosinaemia (TYR) are rare inherited metabolic disorders of amino acid metabolism requiring dietary management. PKU is characterised by an inability to metabolise the essential dietary amino acid phenylalanine (Phe) into tyrosine (Tyr). As such, without appropriate management, PKU can lead to extremely elevated levels of Phe within the blood and brain, which can be detrimental to neurological health. The dietary management of PKU involves restricting dietary sources of Phe. Tyrosinaemia (TYR) is characterised by the inability to metabolise the dietary amino acid Tyr. If left uncontrolled, TYR can lead to serious hepatic, renal and neurological complications. The dietary management of TYR involves restriction of dietary sources of Tyr and Phe (as Phe is converted into Tyr). The dietary management of PKU and TYR involves restricting dietary protein intake to promote optimal metabolic control, whilst meeting all other amino acid and nutrient requirements. As Phe and Tyr are present in significant quantities in nearly all dietary proteins, this usually requires a very low protein diet from food, supplemented with a Phe-free (for PKU) or Phe- and Tyr-free (for TYR) amino acid-based protein substitute. However, compliance with the diet is often poor, with patients commonly going "off diet" during adolescence and in adulthood. This can lead to entirely preventable, lifelong mental and physiological impairments. Reasons for non-compliance often revolve around the strong taste of amino acid-based protein substitutes, alongside the inability to conform to the normal eating habits of peers.

Three new protein substitutes have been developed to help with compliance in PKU and TYR patients, which are powdered protein substitutes, low in Phe and, low in Phe and Tyr respectively, with a mixed balance of glycomacropeptide (GMP), essential and non-essential amino acids, carbohydrates, fats and micronutrients for the dietary management of PKU and TYR. The protein in GMP-based products for PKU and TYR are based on GMP, a peptide isolated from milk during cheese manufacturing and the only known naturally derived protein source low in Phe and Tyr. The GMP is supplemented with appropriate quantities of other amino acids which are naturally low or not present in GMP, as well as carbohydrates and fats. This differs from traditional formulae which are based wholly on individual, synthetically produced amino acids to provide the source of dietary nitrogen, supplemented with vitamins and minerals. Studies to date have illustrated that PKU patients who replace their regular Phe-free amino acid-based formula with GMP-based foods may have better diet compliance, prefer the taste and may have improved blood Phe control.

This series of case-studies will evaluate the acceptability, compliance, gastrointestinal tolerance and safety of the three GMP-based products for PKU and TYR in 45 patients with PKU and TYR, in both adults and children over 3 years (15 patients per product). The case study will last 29 days in total, including a 1-day baseline period followed by a 28-day intervention period. The case studies will be conducted across multiple specialist metabolic centres in the UK, to meet the UK ACBS and GMS requirements for acceptability studies. A series of case studies is undertaken due to the rarity of these conditions and the difficulty in recruiting these patients to trials.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Over 3 years of age
* Diagnosed with classical or variant type phenylketonuria, or tyrosinaemia (as appropriate)
* Have been compliant in taking at least one protein substitute, providing at least 10g protein equivalents, for at least 1 month prior to trial commencement
* Have a prescribed daily Phe or Phe and Tyr allowance for PKU or TYR respectively
* Written or electronic informed consent from patient, and/or from parent/caregiver if applicable

Exclusion Criteria:

* Currently prescribed Sapropterin or similar tetrahydrobiopterin based medication
* Pregnant or lactating
* Requiring parenteral nutrition
* Major hepatic or renal dysfunction
* Participation in other studies within 1 month prior to entry of this study
* Allergy to any of the study product ingredients, including milk and soy
* Investigator concern around willingness/ability of patient or parent/caregiver to comply with protocol requirements

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2020-09-16 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-11-24 (Actual)

PRIMARY OUTCOMES:
Acceptability | Baseline (Day 1) - End of case studies (Day 29)
  Acceptability of the patients' usual protein substitute and the study product assessed by the Dietitian with a series of questions posed to the patient and/or parent/caregiver on on all attributes which included appearance, smell, taste, texture (mouthfeel), ease of mixing, ease of taking, after taste and smell of breath after taking, assessed on a 5-point likert scale (Great; Good; OK; Bad; Terrible).

SECONDARY OUTCOMES:
Compliance | Baseline (Day 1) - End of case studies (Day 29)
  Compliance (% intake compared to that prescribed) with the recommended intake of the patients' usual protein substitute (during baseline) and with the case study product (during the case study period) will be assessed by the Dietitian.
Gastro-intestinal (GI) tolerance | Baseline (Day 1) - End of case studies (Day 29)
  Gastro-intestinal (GI) tolerance symptoms will be recorded by the Dietitian.
Anthropometry | Baseline (Day 1) - End of case studies (Day 29)
  Body weight (kg) and height (m) will be measured where possible using standard methods to calculate body mass index (BMI)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Stratton, Study Chair — Nutricia UK Ltd
Locations (1):
- Bristol University Hospitals, Bristol, United Kingdom

IPD SHARING:
Plan to Share IPD: No